CLINICAL TRIAL: NCT05226767
Title: A Phase II, Randomized, Double-blind, Placebo Controlled Clinical Study Designed to Evaluate the Effect of Daily Oral Administration of Food Supplement NLC-V in Patients Diagnosed With COVID-19
Brief Title: Effect of Daily Oral Administration of Food Supplement NLC-V in Patients Diagnosed With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Todos Medical, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLC-V-01
Record Dates: First submitted 2022-02-01; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: Coronavirus; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Patients who receive treatment with the NLC-V research product depending on the weight of the patients, as follows - Patients weighing less than 70 kg will receive 2 capsules, 4 times a day (80 mg in total per day) Patients weighing between 70 kg and 100 Kg will receive 3 capsules, 4 times a day (a total of 120 mg per day). Patients weighing over 100 kg will receive 4 capsules, 4 times a day (a total of 160 mg per day). NLC-V capsules Will be taken during days 1-10 for the patient's hospitalization NLC-V capsules will be taken during days 1-10 for the patient's hospitalization
  Patients who receive placebo in addition to the usual treatment for COVID-19. The placebo consists of the same solvent, but without the active ingredients of NLC-V. Placebo will be given to patients in the same manner and with the same frequency as NLC-V
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned a 1: 1 ratio to receive NLC-V or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Active Comparator): Patients who receive treatment with the NLC-V research product depending on the weight of the patients, as follows - Patients weighing less than 70 kg will receive 2 capsules, 4 times a day (80 mg in total per day) Patients weighing between 70 kg and 100 Kg will receive 3 capsules, 4 times a day (a total of 120 mg per day). Patients weighing over 100 kg will receive 4 capsules, 4 times a day (a total of 160 mg per day). NLC-V capsules Will be taken during days 1-10 for the patient's hospitalization NLC-V capsules will be taken during days 1-10 for the patient's hospitalization
  Interventions: Dietary Supplement: NLC-V
- Placebo (Placebo Comparator): Patients who receive placebo in addition to the usual treatment for COVID-19. The placebo consists of the same solvent, but without the active ingredients of NLC-V. Placebo will be given to patients in the same manner and with the same frequency as NLC-V
  Interventions: Dietary Supplement: NLC-V

INTERVENTIONS:
Dietary Supplement: NLC-V — NLC-V

SUMMARY:
This study is designed to evaluate the safety and efficacy of NLC-V in patients diagnosed with COVID-19.

DETAILED DESCRIPTION:
Herbal remedies and purified natural products provide a rich resource for the development of new antiviral drugs. The detection of antiviral mechanisms in these natural substances sheds light on where they interact with the viral life cycle, such as penetration, replication, assembly and release of the virus, as well as on tuning to specific host-virus interactions. CoV is a virus that belongs to the corona virus family. The CoV virus family causes infections in the upper respiratory tract and gastrointestinal tract in mammals and birds. In humans, it mainly causes colds, but complications can also occur, such as pneumonia and severe acute respiratory syndrome. Corona virus with the known acute respiratory syndrome caused a global threat with high mortality in 2003, and again in 2019 and 2020.

The plant family of lithosperm, have been used in traditional Chinese medicine for the treatment of external wounds, burns or dermatitis for centuries. Studies conducted over the past 30 years have shown that there is a scientific basis and pharmacological properties. The active ingredients that were successfully extracted from the plant were found to be strong inhibitors of the enzyme family found in corona virus polypropylene 3C. Aim of the study: This study was designed to evaluate the efficacy of NLC-V in patients diagnosed with COVID-19.

Details of the research and clinical follow-up phases: A total of 66 adult patients with a certified diagnosis of SARS-CoV-2 virus infection, who are hospitalized due to the infection, will be recruited. NLC-V study therapy is given in oral capsules. Each NLC-V capsule contains 100 mg of active ingredients in a special formulation. Patients will be randomly assigned a 1: 1 ratio to receive NLC-V or placebo, which are additionally given.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women aged 18 (inclusive) and above.
2. Confirmed SARS-CoV-2 infection by RT-PCR If confirmed >5 days before the randomization, another test will be taken on day 1.
3. Hospitalized COVID-19 patient in stable moderate condition to upper scale of severe condition (i.e., not requiring full respiratory assessment).
4. Oxygenation < 96% on room air.
5. Subjects must be under observation or admitted to a controlled facility or hospital due to lung infection / respiratory infection only (home quarantine is not sufficient).

   -

Exclusion Criteria:

1. Tube feeding or parenteral nutrition.
2. Respiratory decompensation requiring mechanical ventilation.
3. Pregnant or lactating women.
4. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints (for examples social condition other non-related medical illness).
5. Known to have severe allergic reactions to one of the study drug components.
6. Active tuberculosis (TB) infection.
7. Subjects diagnosed to suffer from concomitant active infection: bacterial, fungal, viral, or other infection cause besides COVID-19.
8. In the opinion of the investigator, progression to death is imminent and inevitable within the next 24-36 hours, irrespective of the provision of treatments.
9. Treatment with immunosuppressive or immunomodulatory therapy (including tocilizumab) within the past 3 months (steroids are permitted).
10. Participating in other drug clinical trial.
11. Estimated glomerular filtration rate (eGFR) < 30 mL/min (including patients receiving hemodialysis or hemofiltration).
12. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN) detected within 24 hours of screening (according to local laboratory reference ranges).
13. Absolute neutrophil count (ANC) < 1000/uL at screening.
14. Platelet count < 50,000/uL at screening.
15. Body weight < 40 kg or >120 kg.
16. Treatment with other investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Time relapsed from hospitalization (1st day) until hospital discharge in patients receiving NLC-V treatment. | Time relapsed from hospitalization (1st day) until hospital discharge in patients receiving NLC-V treatment.
Time to clinical improvement, defined as a national Early Warning Score 2 (NEWS2) of </= 2 maintained for 24 hours, in the treatment group (NLC-V) compared to the control group. | Time to clinical improvement, defined as a national Early Warning Score 2 (NEWS2) of </= 2 maintained for 24 hours, in the treatment group (NLC-V) compared to the control group.

SECONDARY OUTCOMES:
Rate of change of measured parameters. | Time relapsed from hospitalization (1st day) until hospital discharge
Rate of change in vital signs (blood pressure, heart rate, respiratory rate, saturation, body temperature). | Time relapsed from hospitalization (1st day) until hospital discharge
Time from the 1st day of receiving NLC-V treatment to negative test result by RT-PCR for COVID-19. | Time relapsed from hospitalization (1st day) until hospital discharge
COVID-19 - related death in the treatment group (NLC-V) compared to the control group. | Time relapsed from hospitalization (1st day) until hospital discharge
Incidence of deterioration and need to mechanical ventilation in both treatment group (NLC-V) and control group. | Time relapsed from hospitalization (1st day) until hospital discharge
Incidence and duration of time on supplemental oxygen in both treatment group (NLC-V) and control group. | Time relapsed from hospitalization (1st day) until hospital discharge
Sensitivity and specificity of NLC's COVID-19 diagnostic test | Time relapsed from hospitalization (1st day) until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Arad, PhD, Study Chair — Todos Medical
Locations (1):
- Shaare Zedek Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No